CLINICAL TRIAL: NCT05756712
Title: A Randomized, Double-blind, Cross-over Clinical Trial of the Efficacy of White Kidney Bean on Oral Glucose Tolerance Test
Brief Title: The Efficacy of White Kidney Bean on Oral Glucose Tolerance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-SM-02-WL-001
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Sugar; Blood, High
Keywords: White Kidney Bean; Oral Glucose Tolerance Test
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wonderlab Product plus Placebo (Active Comparator): Wonderlab product: White Kidney Bean Pressed Candy, 4g/tablet, per serving 750mg extracts of the white kidney bean.
  Placebo: 4g/tablet, per serving 750mg Maltodextrin
  Interventions: Dietary Supplement: Phase 1 Wonderlab Product; Dietary Supplement: Phase 1 Placebo
- Placebo plus Wonderlab Product (Active Comparator): Placebo: 4g/tablet, per serving 750mg Maltodextrin Wonderlab product: White Kidney Bean Pressed Candy, 4g/tablet, per serving 750mg extracts of the white kidney bean.
  Interventions: Dietary Supplement: Phase 2 Placebo; Dietary Supplement: Phase 2 Wonderlab Product

INTERVENTIONS:
Dietary Supplement: Phase 1 Wonderlab Product — Chew two tablets of Wonderlab Product for phase 1 (day 1)
  Arms: Wonderlab Product plus Placebo
Dietary Supplement: Phase 1 Placebo — Washout 72 hours and chew two tablets of placebo for phase 2 (day 4).
  Arms: Wonderlab Product plus Placebo
Dietary Supplement: Phase 2 Placebo — Chew two tablets of placebo for phase 1 (day 1)
  Arms: Placebo plus Wonderlab Product
Dietary Supplement: Phase 2 Wonderlab Product — Washout 72 hours and chew two tablets of Wonderlab Product for phase 2 (day 4).
  Arms: Placebo plus Wonderlab Product

SUMMARY:
The goal of this randomized, double-blind, cross-over inverventional study is to evaluate the efficacy of white kidney bean on OGTT (oral glucose tolerance test). About 34 eligible participants will be randomized in two groups of the same size to take the assigned interventions at one study site in Shanghai, two visits will be required. The first group of participants will take Wonderlab product first and then placebo product after 72 hours of washout period, while the other group of of participants will take placebo product first and then Wonderlab product after 72 hours of washout period. For each visit, the finger blood will be sampled and the relevent data such as blood glucose will be captured based on OGTT procedures, and recorded into clinical data management system for statistical analysis.

Researchers will compare the two groups to see if there is significant change of blood glucose by using products containing ingredient of white kidney beans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 25-45 years, with a male to female ratio of more than 40% and BMI 24.

  35 subjects enrolled and 30 subjects completed the study;
* There is no history of diabetes and other metabolic syndrome, digestive diseases, endocrine disorder and mental diseases;
* No history of food allergy and intolerance;
* No nutritional supplements that affect glucose tolerance, oral contraceptives, acetylsalicylic acid, steroids, protease inhibitors, and antipsychotic drugs in the past 3 months;
* Able to tolerate at least 10 hours of fasting;
* Willing to refrain from participating in other interventional clinical studies during the trial period;
* Be able to fully understand the purpose, benefits and potential risks including side effects of the research;
* Willing to obey all test requirements and procedures;
* Informed consent signed.

Exclusion Criteria:

* Subject who is in the treatment of gastrointestinal diseases;
* Subjects are currently suffering from other organic diseases that affect intestinal function, such as history of gastrointestinal resection, colonic or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, Hirschsprung's disease, scleroderma, anorexia nervosa, etc.;
* Controlling diet, exercising, or taking medications to control weight or affect appetite in the last 3 months;
* Subjects have any of the following medical history or have been clinically examined to have the following diseases that may affect the evaluation of the test effect: obvious gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases;
* Abuse alcohol or other drugs, supplement or OTC drugs currently or n the past may cause bowel dysfunction or can affect test result evaluation;
* Frequently use of medications that may affect gastrointestinal function or the immune system according to investigator's judgment;
* Take laxatives or other substances that promote digestion 2 weeks before the trail start;
* Pregnant or lactating women or those planning to become pregnant during the trial;
* Liver function tests (alanine aminotransferase and aspartate aminotransferase), renal function tests (blood urea nitrogen and creatinine), routine blood tests, urinalysis, fecal occult blood test or electrocardiogram abnormalities.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The Change of Blood Glucose Level in mmol/L based on OGTT (Oral Glucose Tolerance Test) after Intervention | At the end of Phase 1 and Phase 2 (each phase is 1 day)
  The Change of Blood Glucose Level in mmol/L based on OGTT (Oral Glucose Tolerance Test) after intervention: Chewing Wonderlab Product - White Kidney Bean Pressed Candy, followed by Placebo Product at the interval of washout duration of 72 hours; and Chewing Placebo Product, followed by Wonderlab Product - White Kidney Bean Pressed Candy at the interval of washout duration of 72 hours.

SECONDARY OUTCOMES:
The Change of Fast Blood Glucose Level in mmol/L based on OGTT (Oral Glucose Tolerance Test) after Intervention | At the end of Phase 1 and Phase 2 (each phase is 1 day)
  The Change of Fast Blood Glucose Level in mmol/L based on OGTT (Oral Glucose Tolerance Test) after intervention: Chewing Wonderlab Product - White Kidney Bean Pressed Candy, followed by Placebo Product at the interval of washout duration of 72 hours; and Chewing Placebo Product, followed by Wonderlab Product - White Kidney Bean Pressed Candy at the interval of washout duration of 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — SPRIM Medical
Locations (1):
- SPRIM Central Lab, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No